CLINICAL TRIAL: NCT06969625
Title: Shoulder Anterior Capsular Block Versus Combined Suprascapular and Axillary Nerve Blocks for Postoperative Analgesia in Arthroscopic Rotator Cuff Repair Surgery
Brief Title: Shoulder Anterior Capsular Block for Postoperative Analgesia in Arthroscopic Rotator Cuff Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Associate professor of anaesthesia, intensive care, and pain management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1271/27-4-2025
Record Dates: First submitted 2025-05-03; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Arthroscopic Rotator Cuff Repair
Keywords: shoulder anterior capsular block; combined suprascapular and axillary nerve blocks; postoperative analgesia; arthroscopic rotator cuff repair surgery
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (SHAC) block (Experimental)
  Interventions: Procedure: (SHAC) block
- Group (SSNB-ANB) block (Active Comparator)
  Interventions: Procedure: (SSNB-ANB) block

INTERVENTIONS:
Procedure: (SHAC) block — The shoulder anterior capsular block targets interfacial and pericapsular space. A 25-gauge 80-mm insulated stimulating needle will be used for injections and in-plane needling will be from lateral to medial side. After aspiration is negative, 10 ml of 0.5 % bupivacaine plus dexamethasone 4 mg as adjuvant will be injected in the interfacial plane. Once the injection into the fascial space is achieved, the operator can proceed towards the glenohumeral pericapsular space by crossing the subscapularis muscle with the needle and the second injection after negative aspiration will be 10 ml 0.5 % bupivacaine plus dexamethasone 4 mg in pericapsular space.
  Arms: Group (SHAC) block
Procedure: (SSNB-ANB) block — Suprascapular Nerve Block (SNB): Using an in-plane ultrasound guidance from the medial side, 10 mL of 0.5% bupivacaine plus dexamethasone 4 mg as adjuvant will be injected after contacting the lateral aspect of the supraspinous fossa and negative aspiration confirmed. The LA should spread beneath the supraspinatus, lifting up the muscle.
  Axillary Nerve Block (ANB):
  The ANB is performed from behind the patient with the patient seated. The axillary nerve will be identified within the quadrilateral space by placing high frequency linear probe (Sono site M turbo) parallel to the long axis of the humeral shaft. The nerve was identified next to the circumflex artery. The skin will be anesthetized with 1% lidocaine (3mL). 10 mL of 0.5% bupivacaine plus dexamethasone 4 mg will be injected against the surface of the humerus, just posterior and lateral to the artery after confirming negative aspiration.
  Arms: Group (SSNB-ANB) block

SUMMARY:
Shoulder pain is frequently encountered in the medical field. Rotator cuff tears are the most common cause. Shoulder pain affects quality of life and delay rehabilitation programs.

Effective control of post operative pain is a cornerstone in the success of these surgeries. Regional anaesthesia is often favoured for shoulder surgery as it could effectively provide anaesthesia and postoperative analgesia. Additionally, the upper limb has multiple nerve targets that can be blocked. Ultrasound combined SSNB-ANB were described as an alternative to interscalene nerve block for shoulder surgeries equipotent pain relief and patient satisfaction as well as fewer complications due to the location of injection.

Ultrasound guided SHAC block is a motor sparing block which targets all nerves supplying shoulder consistently at two sites. It was validated in chronic shoulder pain patients. However, there is no sufficient evidence for this block in postoperative pain after shoulder surgery.

DETAILED DESCRIPTION:
Regional anaesthesia is often favoured for shoulder surgery as it could effectively provide anaesthesia and postoperative analgesia. Additionally, the upper limb has multiple nerve targets that can be blocked. Innervation of shoulder joint is complex with 70 % contribution from suprascapular nerve (SSN), remaining from axillary (AN), lateral pectoral, subscapular, and musculocutaneous nerves. Therefore, Effective postoperative analgesia for shoulder surgery should target mainly both the SSN and AN which can be performed either at the level of the nerves themselves or their more proximal origins, often within the brachial plexus.

Until recently, interscalene brachial plexus block (ISB) was considered the gold standard technique for intra- and postoperative pain management in shoulder surgeries. However, its safety was questioned due to its drawbacks including prolonged motor block, and most importantly hemidiaphragm paralysis and the resultant pulmonary function compromise with prolongation of the patients' recovery time. The shoulder block which refers to the combined suprascapular nerve and axillary nerve block (SSNB-ANB) was first described in 2007 as an alternative to interscalene block (ISB) for shoulder surgeries with several studies reporting equipotent pain relief and patient satisfaction when the combined SSNB -ANB compared with the ISB alone with fewer complications due to the location of injection.

In 2020, Galluccio et al. described a novel ultrasound-guided block, the shoulder anterior capsular block (SHAC), motor sparing block, which blocks all the nerves supplying the shoulder based on the combination of two blocks targeting the interfacial and pericapsular spaces. Thanks to this approach which block axillary, subscapular, lateral pectoral and musculocutaneous nerves and avoid motor block associated with more proximal nerve blocks, thus allowing early active mobilization, physiotherapy and rehabilitation.

SHAC block was validated in chronic shoulder pain patients. hence, we hypothesized that SHAC block is effective in postoperative shoulder pain relief and early rehabilitation after ARCR which could make it an alternative to SSNB-ANB in these patients. This study will be undertaken to compare between the analgesic effect of ultrasound guided SHAC block versus combined ultrasound guided SSNB-ANB for arthroscopic rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients acceptance
* Age: 21-60 years
* Sex: both sexes (males or females).
* Physical status: ASA 1& II.
* Body mass index (BMI) ≤ 30 kg/m2
* Type of operation: arthroscopic rotator cuff repair surgery.
* Duration of surgery: within 2 hours.

Exclusion Criteria:

* Patient with any contraindications of regional blocks (as coagulopathy or local infection at injection site)
* Patients with known history of allergy to the study drugs.
* patients with neuropathy involving the limb undergoing surgery
* Advanced hepatic, renal, cardiovascular, and neurologic diseases.
* history of previous shoulder operation or fracture.
* conversion to open surgery from arthroscopy.
* pregnant females
* patients with chronic opioid use

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The total postoperative pethidine consumption (in milligrams) during the first 24-h after surgery. | 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain assessment by Numeric rating scale (NRS) at rest and on passive movements in the recovery room and at 2,4,8,16 and 24 hours after surgery. | 24 hours after surgery
  The patients will be instructed to use numeric rating scale (NRS) for pain. The numeric rating scale will be explained using a 0-10 scale, with the left-most end (zero) meaning "no pain" and the right-most end (10) meaning "the worst pain imaginable". Patients will be instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation
The time to first request of rescue analgesia (pethidine). | 24 hours after surgery
3. The total number of patients requiring additional dose of intraoperative fentanyl. | 3 hours
The block performance time | 1 hour
  defined by the sum of scanning time and needle time. Scanning time is the time from ultrasound probe is placed on the skin until a satisfactory image is obtained. Needle time is taken from the time needle tip penetrated the skin and exited after block placement.
Over all patients' satisfaction on the next day of surgery | 24 hours after surgery
  by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia).
The incidence of any complications | 7 days after surgery
  block related complications including hematoma, local anesthetic toxicity, infection, persistent paresthesia, weakness, and tingling at 1 and 7 days after surgery - opioid related side effects including nausea, vomiting, and sedation).

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E. Abd Ellatif, MD, Study Director — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University; Sherif M. S. Mowafy, MD, Principal Investigator — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University; Fatma M. Ahmed, MD, Study Chair — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: from the study director

REFERENCES:
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Galluccio F, Fajardo Perez M, Yamak Altinpulluk E, Hou JD, Lin JA. Evaluation of Interfascial Plane and Pericapsular Nerve Blocks to the Shoulder Joint: A Preliminary Analysis of Shoulder Anterior Capsular Block. Pain Ther. 2021 Dec;10(2):1741-1754. doi: 10.1007/s40122-021-00326-0. Epub 2021 Oct 20. PMID 34669181
- [Background] Galluccio F, Arnay EG, Salazar C, Altinpulluk EY, Capassoni M, Garcia DS, Espinoza K, Olea MS, Perez MF. Re: "Ultrasound-Guided Block of the Axillary Nerve: A Prospective, Randomized, Single-Blind Study Comparing Interfascial and Perivascular Injections". Pain Physician. 2020 Jan;23(1):E62-E64. No abstract available. PMID 32013290
- [Background] Zhao J, Xu N, Li J, Liang G, Zeng L, Luo M, Pan J, Yang W, Liu J. Efficacy and safety of suprascapular nerve block combined with axillary nerve block for arthroscopic shoulder surgery: A systematic review and meta-analysis of randomized controlled trials. Int J Surg. 2021 Oct;94:106111. doi: 10.1016/j.ijsu.2021.106111. Epub 2021 Sep 11. PMID 34520842
- [Background] Faiz SHR, Mohseni M, Imani F, Attaee MK, Movassaghi S, Rahimzadeh P. Comparison of Ultrasound-Guided Supra-scapular Plus Axillary Nerve Block with Interscalene Block for Postoperative Pain Management in Arthroscopic Shoulder Surgery; A Double-Blinded Randomized Open-Label Clinical Trial. Anesth Pain Med. 2021 May 2;11(2):e112540. doi: 10.5812/aapm.112540. eCollection 2021 Apr. PMID 34336619
- [Background] Price DJ. The shoulder block: a new alternative to interscalene brachial plexus blockade for the control of postoperative shoulder pain. Anaesth Intensive Care. 2007 Aug;35(4):575-81. doi: 10.1177/0310057X0703500418. PMID 18020078
- [Background] Divella M, Vetrugno L, Orso D, Langiano N, Bignami E, Bove T, Della Rocca G. Interscalenic versus suprascapular nerve block: can the type of block influence short- and long-term outcomes? An observational study. Minerva Anestesiol. 2019 Apr;85(4):344-350. doi: 10.23736/S0375-9393.18.12791-X. Epub 2018 Jul 9. PMID 29991222
- [Background] Brull R, McCartney CJ, Chan VW, El-Beheiry H. Neurological complications after regional anesthesia: contemporary estimates of risk. Anesth Analg. 2007 Apr;104(4):965-74. doi: 10.1213/01.ane.0000258740.17193.ec. PMID 17377115
- [Background] Lim YC, Koo ZK, Ho VW, Chang SS, Manohara S, Tong QJ. Randomized, controlled trial comparing respiratory and analgesic effects of interscalene, anterior suprascapular, and posterior suprascapular nerve blocks for arthroscopic shoulder surgery. Korean J Anesthesiol. 2020 Oct;73(5):408-416. doi: 10.4097/kja.20141. Epub 2020 Jul 16. PMID 32668833
- [Background] Rhyner P, Kirkham K, Hirotsu C, Farron A, Albrecht E. A randomised controlled trial of shoulder block vs. interscalene brachial plexus block for ventilatory function after shoulder arthroscopy. Anaesthesia. 2020 Apr;75(4):493-498. doi: 10.1111/anae.14957. Epub 2019 Dec 19. PMID 31854463
- [Background] Morita S, Oizumi N, Suenaga N, Yoshioka C, Yamane S, Tanaka Y. Dexamethasone added to levobupivacaine prolongs the duration of interscalene brachial plexus block and decreases rebound pain after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2020 Sep;29(9):1751-1757. doi: 10.1016/j.jse.2020.04.019. Epub 2020 Jun 9. PMID 32815804
- [Background] Shishido H, Kikuchi S, Heckman H, Myers RR. Dexamethasone decreases blood flow in normal nerves and dorsal root ganglia. Spine (Phila Pa 1976). 2002 Mar 15;27(6):581-6. doi: 10.1097/00007632-200203150-00005. PMID 11884905
- [Background] 4. Vaidiyanathan B, Sundaresan S, Raajesh I. "Shoulder Anterior Capsular Block: An Effective Strategy for Alleviating Pain During Shoulder Mobilisation in Adhesive Capsulitis Patients": A Case Series. Arch Anesth & Crit Care. 2024;10(Supp. 1):526-29.
- [Background] Borgeat A, Ekatodramis G. Anaesthesia for shoulder surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):211-25. doi: 10.1053/bean.2002.0234. PMID 12491553
- [Background] Patel MS, Abboud JA, Sethi PM. Perioperative pain management for shoulder surgery: evolving techniques. J Shoulder Elbow Surg. 2020 Nov;29(11):e416-e433. doi: 10.1016/j.jse.2020.04.049. Epub 2020 Jun 9. PMID 32844751
- [Background] Blom AW, Donovan RL, Beswick AD, Whitehouse MR, Kunutsor SK. Common elective orthopaedic procedures and their clinical effectiveness: umbrella review of level 1 evidence. BMJ. 2021 Jul 7;374:n1511. doi: 10.1136/bmj.n1511. PMID 34233885